CLINICAL TRIAL: NCT06119555
Title: Investigating the Impact of Consuming Cinnamon Powder on the Body Composition Among Obese University Students in Lahore
Brief Title: Effect of Cinnamon Powder Capsules on Body Composition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Muhammad Shahbaz, Associate Professor, Department of Food Sciences and Human Nutrition, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cinnamon Bark Powder Capsules
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Body Composition
Keywords: Obesity; Cinnamon; Body Mass Index; Body Fat Mass; Percent Body Fat; Skeletal Muscle Mass; Waist-to-hip Ratio
MeSH Terms: conditions — Obesity | interventions — camphorin protein, Cinnamomum camphora

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon Group (Experimental): In the cinnamon group, participants will consume four cinnamon capsules daily for 60 days (each 1.5 grams, totaling 3 grams), two with breakfast and two with dinner.
  Interventions: Dietary Supplement: Cinnamon Capsules
- Control Group (No Intervention): The control group will not receive intervention.

INTERVENTIONS:
Dietary Supplement: Cinnamon Capsules — The intervention consists of four cinnamon capsules (each 1.5 grams, totaling 3 grams) a day, with two with breakfast and two with dinner for 60 days
  Other Names: Cinnamomum; Dalchini; Darchini
  Arms: Cinnamon Group

SUMMARY:
Obesity is a global health concern that significantly affects individuals, and its prevalence is still rising at an alarming rate. While various treatments are available, they often come with unwanted side effects. As a result, there is a growing interest in natural remedies including various herbs and spices such as cinnamon that have a favorable impact on overall health and disease conditions.

DETAILED DESCRIPTION:
Obesity is a global health concern that significantly affects individuals, and its prevalence is still rising at an alarming rate. Pakistan is also experiencing an increasing prevalence of obesity, resulting in elevated morbidity, mortality, and healthcare costs. While various treatments are available, they often come with negative side effects that can reduce a patient's quality of life. Correspondingly, natural remedies have a kindle appeal that can enhance overall health and well-being. In Pakistani culture, natural condiments have been used for their health and therapeutic benefits. Cinnamon, an ancient spice commonly found in various regions, contains active ingredients that offer several health benefits. However, there is limited scientific data regarding the effects of cinnamon on body composition, especially among obese university students in Pakistan. Therefore, the current study aims to investigate the potential outcome of orally consuming cinnamon for weight management in obese university students in Pakistan. As a result, the study may provide effective evidence-based strategies for maintaining healthy body weight and exploring the potential use of cinnamon as a natural treatment option.

ELIGIBILITY:
Inclusion Criteria:

* Obese individuals (≥ 25 kg/m^2)
* University students of all disciplines
* Participants of 18-28 years
* Both male and female

Exclusion Criteria:

* Morbid obesity (BMI ≥30 kg/m^2)
* Disease conditions (such as cardiovascular diseases, diabetes, hypertension, renal disease, hypothyroidism, and hyperthyroidism)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Waist-to-hip ratio | 60 days
  The waist-to-hip ratio will be assessment before and after intervention with cinnamon powder capsules for 60 days.
Body weight | 60 days
  Body weight (Kg) will be assessed before and after intervention with cinnamon powder capsules for 60 days.
Skeletal muscle mass (SMM) | 60 days
  Skeletal muscle mass (Kg) will be assessed before and after intervention with cinnamon powder capsules for 60 days.
Body fat mass | 60 days
  Body fat mass (Kg) will be assessed before and after intervention with cinnamon powder capsules for 60 days.
Body mass index (BMI) | 60 days
  Body mass index (Kg/m^2) will be assessed before and after intervention with cinnamon powder capsules for 60 days.
Percent body fat (PBF) | 60 days
  Percent body fat (%) will be assessed before and after intervention with cinnamon powder capsules for 60 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Veterinary and Animal Sciences, Lahore - Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
All available data will be confidential

REFERENCES:
- [Result] Gupta Jain S, Puri S, Misra A, Gulati S, Mani K. Effect of oral cinnamon intervention on metabolic profile and body composition of Asian Indians with metabolic syndrome: a randomized double -blind control trial. Lipids Health Dis. 2017 Jun 12;16(1):113. doi: 10.1186/s12944-017-0504-8. PMID 28606084
- See also: Oral cinnamon intervention improves metabolic profile and body composition of individuals with metabolic syndrome — http://pubmed.ncbi.nlm.nih.gov/28606084/